CLINICAL TRIAL: NCT02801279
Title: Development of Kinect-assisted Home-based Bilateral Arm Training Program for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201503112RIND
Record Dates: First submitted 2016-06-13; First posted 2016-06-15 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Occupational Therapy; Upper Limb Motor Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinect-based bilateral arm training (Experimental): The Kinect-based bilateral arm training focuses activities that required the use of both hands by using Kinect game.
  Interventions: Other: Kinect-based bilateral arm training
- Conventional bilateral arm training (Experimental): The conventional bilateral arm training focuses activities that required the use of both hands.
  Interventions: Other: Conventional bilateral arm training

INTERVENTIONS:
Other: Conventional bilateral arm training — The Kinect-based bilateral arm training focuses activities that required the use of both hands by using Kinect game.
  Arms: Conventional bilateral arm training
Other: Kinect-based bilateral arm training — The conventional bilateral arm training focuses activities that required the use of both hands.
  Arms: Kinect-based bilateral arm training

SUMMARY:
The purpose of the present study is to develop a long term cost-effectiveness (efficient protocol, playful context, and practical strategy) training program for school-age children with Cerebral Palsy. Also, evaluate efficacy of Kinect-assisted bilateral arm training program for children with Cerebral Palsy.

ELIGIBILITY:
The inclusion criteria of children with CP are:

1. diagnosed with congenital hemiplegic
2. no excessive muscle tone (Modified Ashworth Scale ≤ 3 at any joints of the upper limb)

The exclusion criteria of children with CP are:

1. have severe cognitive, visual, or auditory disorders according to medical documents, parental reports, and the examiner's clinical observation
2. have injections of botulinum toxin type A.

The inclusion criteria of typically developing children are:

1. absence of medical or developmental diseases which would affect physical and cognitive performances
2. having normal corrected vision
3. studying in regular education classroom in primary school for the 6-12 year-old children.

The exclusion criteria of typically developing children are:

(1) having score not within normal limits in BOTMP-short form

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Performance change of Kinematic analysis | baseline, after 8 weeks, after 6 months

SECONDARY OUTCOMES:
Change of muscle strength | baseline, after 8 weeks, after 6 months
Score change of Melbourne Assessment 2 (MA-2) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Pediatric Motor Activity Log-Revised (PMAL-R) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of ABILHAND-Kids | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Test of Playfulness (ToP) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Box and Block Test (BBT) | baseline, every week(week1 to week 8), after 4 weeks, after 8 weeks, after 6 months
Score change of Engagement Questionnaire (EQ) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Satisfactory Questionnaire (SQ) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Building Tower Test (BTT) | baseline, every week(week1 to week 8), after 4 weeks, after 8 weeks, after 6 months
Score change of String Beads Test (SBT) | baseline, every week(week1 to week 8), after 4 weeks, after 8 weeks, after 6 months
Score change of Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Pediatric Evaluation of Disability Inventory (PEDI) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Cerebral Palsy Quality of Life Questionnaire for Children (CPQOL) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Parenting Stress Index-Short Form (PSI-short) | baseline, after 4 weeks, after 8 weeks, after 6 months
Score change of Test of Visual Perceptual Skills | baseline, after 4 weeks, after 8 weeks, after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Ling Chen, Principal Investigator — Taiwan University, Department of Occupational Therapy
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan